CLINICAL TRIAL: NCT06767761
Title: A Phase III Clinical Study Comparing the Efficacy and Safety of Once-weekly GZR4 Versus Once-daily Insulin Glargine U100 in Combination With Insulin Aspart (With or Without Non-Insulin Antidiabetic Agents) in Subjects With Type 2 Diabetes Mellitus (T2DM) Treated With Basal+Prandial Insulin Treatment
Brief Title: A Phase III Clinical Study to Assess the Efficacy and Safety of GZR4 in Type 2 Diabetes Mellitus Subjects (T2DM) Treated With Basal + Prandial Insulin
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR4-T2D-303
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Diabetes
Keywords: GZR4; insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR4 group (Experimental)
  Interventions: Drug: GZR4
- Insulin Glargine U100 group (Active Comparator)
  Interventions: Drug: Insulin Glargine U100 group

INTERVENTIONS:
Drug: GZR4 — GZR4 s.c., once-weekly，treat-to-target dose
  Arms: GZR4 group
Drug: Insulin Glargine U100 group — Insulin Glargine U100 s.c.,once-daily，treat-to-target dose
  Arms: Insulin Glargine U100 group

SUMMARY:
This study will be conducted to compare the efficacy, safety and patient-reported outcome of once-weekly GZR4 and once-daily Insulin Glargine U100 in Combination with Insulin Aspart (with or without Non-Insulin Antidiabetic Agents) in Subjects with Type 2 Diabetes Mellitus (T2DM) Treated with Basal+Prandial Insulin Treatment

ELIGIBILITY:
Inclusion Criteria:

* Sign the Informed Consent Form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and be able to follow the contraindications and restrictions specified in this protocol.
* Males and females age ≥ 18 years at the time of informed consent.
* The pregnancy test for β-human chorionic gonadotropin (hCG) must be negative for women of childbearing potential during the screening period and prior to randomization.
* From signing the Informed Consent Form until 3 weeks after the end of treatment, female subjects of childbearing potential and male subjects and their partners must agree to use reliable contraceptive measures and not donate eggs (ova, oocytes) or sperm for assisted reproductive purposes.
* According to the diagnostic criteria and classification of diabetes mellitus issued by the World Health Organization (WHO) in 1999, and the supplementary diagnostic criteria recommended by WHO for diagnosis with Hemoglobin A1c (HbA1c) (2011), the time to diagnose T2DM is ≥ 180 days at screening.
* Prior to screening, one basal insulin once daily and prandial insulin 2 ~ 4 times daily was given. Or 1 or 2 times daily of a premixed insulin analogue or dual insulin analogue.

Exclusion Criteria:

* A history of allergy to drugs with two or more mechanisms of action in the past, or known allergies, hypersensitivity, or intolerance to the investigational medicinal product or its excipients (glycerol, phenol, m-cresol, zinc acetate dihydrate, sodium chloride, citric acid monohydrate, or zinc chloride).
* Subjects who are pregnant, lactating or planning to become pregnant during the study at screening.
* Participated in any drug clinical study (received non-placebo medication during the study) within a recent period of time (90 days or 5 half-lives of the previous investigational medicinal product, whichever is longer), or plans to participate in another clinical study before completing all scheduled assessments in this clinical study.
* Underwent invasive cardiovascular or cerebrovascular procedures within 180 days before screening; or experienced acute heart failure, myocardial infarction, stroke, or hospitalization due to angina unstable, transient ischaemic attack, or other acute cardiovascular events within 180 days before screening; or have a history of chronic cardiac failure classified as New York Heart Association Class III or IV at screening; or plan to undergo coronary, carotid, or peripheral arterial revascularisation procedures during the study; or have clinically significant abnormalities on the electrocardiogram (ECG) that require treatment at screening (such as second-degree type II or third-degree atrioventricular block, ventricular fibrillation, ventricular flutter, atrial fibrillation, atrial flutter, Wolff-Parkinson-White syndrome, etc.).
* History of malignant tumors before screening (excluding adequately treated or resected non-metastatic basal or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer in situ) or the presence of underlying malignancy at screening.
* The patient with SBP ≥ 160 mmHg or DBP ≥ 100 mmHg during screening.
* Subjects who are unable to comply with the requirements of this protocol as judged by the investigator, or have any other conditions that the investigator considers inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to week 26

SECONDARY OUTCOMES:
hypoglycaemia events | From baseline (week 0) to week 26
adverse events | From baseline (week 0) to week 26
Change in weight | From baseline (week 0) to week 26

CONTACTS AND LOCATIONS:
Locations (1):
- The Second XIANGYA Hospital Of Central South University, Changsha, Hunan, China